CLINICAL TRIAL: NCT00301795
Title: A Phase II Trial of Rituximab + Oblimersen Sodium (GenasenseTM, G3139, NSC #683428, IND #58842) in Patients With Previously Untreated Follicular Non-Hodgkin Lymphoma (NHL)
Brief Title: Rituximab and Oblimersen in Treating Patients With Stage II, Stage III, or Stage IV Follicular Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03080; CALGB 50404; U10CA031946 (NIH); CDR0000462385 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — oblimersen; Rituximab

ARMS (1):
- Treatment (oblimersen sodium and rituximab) (Experimental): Induction therapy (month 1): Patients receive oblimersen IV continuously on days 1-7 and 15-21 and rituximab IV on days 3, 10, 17, and 24 in month 1.
  Extended induction therapy (months 3, 5, 7, and 9): Patients receive oblimersen IV continuously on days 22-28 and rituximab IV on day 24 in months 3, 5, 7, and 9.
  Treatment continues for 9 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: oblimersen sodium; Biological: rituximab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Oblimersen may help rituximab work better by making cancer cells more sensitive to the drug. This phase II trial is studying how well giving rituximab together with oblimersen works in treating patients with stage II, stage III, or stage IV follicular non-Hodgkin's lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (overall and complete response rate) after rituximab + oblimersen sodium extended induction therapy in previously untreated cluster of differentiation 20 positive (CD20+) follicular non-Hodgkin lymphoma (NHL) patients.

II. To determine the time to progression after rituximab + oblimersen sodium extended induction therapy in previously untreated CD20+ follicular NHL patients.

SECONDARY OBJECTIVES:

I. To determine the toxicity profile of rituximab + oblimersen sodium therapy in previously untreated CD20+ follicular NHL patients.

II. To establish whether the therapeutic effects of the rituximab + oblimersen sodium combination are sufficiently promising to warrant evaluation in a subsequent randomized trial (in comparison to rituximab alone).

III. To correlate Fc receptor profiling to response to rituximab + oblimersen sodium in previously untreated patients with follicular NHL.

IV. To determine the relationship between change in fludeoxyglucose F 18 (FDG) uptake early after treatment with rituximab + oblimersen sodium to response rate and time to progression.

OUTLINE: This is a multicenter study.

Induction therapy (month 1): Patients receive oblimersen IV continuously on days 1-7 and 15-21 and rituximab IV on days 3, 10, 17, and 24 in month 1.

Extended induction therapy (months 3, 5, 7, and 9): Patients receive oblimersen IV continuously on days 22-28 and rituximab IV on day 24 in months 3, 5, 7, and 9.

Treatment continues for 9 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 52 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed follicular lymphoma, WHO classification, grade 1, 2, or 3a (> 15 centroblasts per high power field with centrocytes present) which is stage III, IV, or bulky (i.e., single mass >= 7 cm in any unidimensional measurement) stage II
* Institutional flow cytometry or immunohistochemistry must confirm CD20 antigen expression
* Patients classified as high risk according to the Follicular Lymphoma International Prognostic Index (FLIPI) should be considered for CALGB 50102/SWOG S0016
* No prior therapy for non-Hodgkin lymphoma including chemotherapy, radiation or immunotherapy (e.g., monoclonal antibody-based therapy)
* No corticosteroids within two weeks prior to study, except for maintenance therapy for a non-malignant disease
* ECOG performance status 0-2
* Measurable disease must be present either on physical examination or imaging studies; non-measurable disease alone is not acceptable; any tumor mass > 1 cm is acceptable; lesions that are considered non-measurable include the following:

  * Bone lesions (lesions if present should be noted)
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Bone marrow (involvement by non-Hodgkin lymphoma should be noted)
* No known CNS involvement by lymphoma
* No known HIV infection
* Non-pregnant and non-nursing; women and men of reproductive potential should agree to use an effective means of birth control throughout their participation in this study; appropriate methods of birth control include oral contraceptives, implantable hormonal contraceptives, or double barrier method (diaphragm plus condom)
* Patients with a "currently active" second malignancy, other than nonmelanoma skin cancers are not eligible; (this includes Waldenstrom's Macroglobulinemia, since such patents have experienced transient increases in IgM following initiation of rituximab, with the potential for hyperviscosity syndrome requiring plasmapheresis); patients are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy, and are considered by their physician to be at less than 30% risk of relapse
* ANC >= 1000/uL
* Platelet count >= 50,000/uL
* Creatinine =< 2 x ULN
* Total bilirubin =< 2 x ULN; unless attributable to Gilbert's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2006-03; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Overall response (OR) rate defined as achievement of a complete (CR) or partial response (PR) as the best observed response | 12 months
  The true OR rate will be estimated using the uniformly minimum unbiased estimator. Jennison and Turnbull's method will be used to obtain 95% exact confidence interval for the true OR rate of each arm reflecting the above two-stage design.

SECONDARY OUTCOMES:
Toxicities assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 10 years
  Will be summarized using frequency tables.
Time-to-progression (TTP) | Up to 10 years
  Kaplan-Meier method will be used.
Time-to-best response | Up to 10 years
  Kaplan-Meier method will be used.
Overall survival | Up to 10 years
  Kaplan-Meier method will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Grant, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States